CLINICAL TRIAL: NCT06343077
Title: Phase II Trial of In-Situ Autologous Vaccination With Intratumoral and Systemic Hiltonol® (Poly-ICLC) Administered to Prostate Cancer Patients on Active Surveillance
Brief Title: Intratumoral and Systemic Hiltonol® (Poly-ICLC) in Prostate Cancer Patients on Active Surveillance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ashutosh Kumar Tewari (Other)
Collaborators: Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ashutosh Kumar Tewari, Professor and System Chair, Milton and Carroll Petrie Department of Urology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-22-00106
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer Patients on Active Surveillance
Keywords: Prostate Cancer; Active Surveillance; Vaccination; Immunotherapy; drug POLY-ICLC; Gleason Grade 2 (Gleason 3+4); Gleason Grade 1 (Gleason 3+3)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections; poly ICLC

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hiltonol (Poly-ICLC) (Active Comparator): Enrolled study subjects will receive paired intramuscular (IM) and intertumoral. (IT) injections of the drug Poly-ICLC (Hiltonol®) as follows: Paired 1.5 mg IM (week 1), 1 mg IT once (week 2), followed by paired 1.5 mg IM weekly from weeks 3-through10, and at weeks 14, 18, 22, 26, 30, 34, 38, 42 and 46 with a 4-week rest period between IM injections.
  Interventions: Drug: Poly-ICLC intramuscular (IM) injection; Drug: Poly-ICLC, Intertumoral (IT) injection
- Control (Standard of Care) (No Intervention)

INTERVENTIONS:
Drug: Poly-ICLC intramuscular (IM) injection — 1.5 mg IM (week 1), followed by paired 1.5 mg IM weekly from weeks 3-through10, and at weeks 14, 18, 22, 26, 30, 34, 38, 42 and 46 with a 4-week rest period between IM injections.
  Other Names: Hiltonol®; Polyinosinic-Polycytidylic acid stabilized with polylysine and carboxymethylcellulose
  Arms: Hiltonol (Poly-ICLC)
Drug: Poly-ICLC, Intertumoral (IT) injection — 1 mg IT once (week 2)
  Other Names: Hiltonol®; Polyinosinic-Polycytidylic acid stabilized with polylysine and carboxymethylcellulose
  Arms: Hiltonol (Poly-ICLC)

SUMMARY:
This is a partially blinded randomized controlled phase II pilot study comparing Poly-ICLC (Hiltonol®) treatment vs no treatment, for prostate cancer participants on active surveillance.

DETAILED DESCRIPTION:
114 prostate cancer participants on active surveillance will be randomized 2:1 into treatment group, A or control group B respectively. Enrolled group A study participants will receive standard of care (SOC) plus intratumoral (IT) and intramuscular (IM) injections of study drug Poly-ICLC (Hiltonol®) as follows:

Preconditioning: week 1: Paired IM Poly-ICLC, 1.5 mg to reduce tumor induced suppression

Immune Priming: week 2, intratumor poly-ICLC 1.0 mg once,

Boosting: Wk. 3 - 10: Paired 1.5 mg IM poly-ICLC weekly

Maintenance: Month 3-12, Paired IM Poly-ICLC once a month

Control patients in group B will receive standard care (SOC) for patients on Active Surveillance per AUS guidelines.

Comparisons of safety and efficacy will be based on data from concurrently randomized participants. An independent data and safety monitoring board (DSMB) will actively monitor interim data for safety, efficacy or futility.

Seventy-six (76) participants will receive treatment IT/IM Poly-ICLC (Hiltonol®) and 38 participants will serve as controls for a total of 114 study participants. Participants randomized to the treatment arm will receive standard of care (SOC) plus IT/IM Poly-ICLC (Hiltonol®). Participants in the control arm will receive SOC. This is a partially blind randomized controlled phase 2 trial conducted at the Mount Sinai Health System with 114 participants planned for enrollment. Eligible participants will be randomly assigned to one of the two groups.

There will be an interim analysis conducted after half of the participants, 38 receiving Poly-ICLC and 19 controls receiving standard care have completed 1 year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.

NOTE: HIPAA authorization may be included in the informed consent or obtained separately.

* Age > 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 14 days prior to being registered for protocol therapy (Study Procedure Manual).
* Histologically confirmed adenocarcinoma of the prostate (with previous diagnostic tissue available for tumor marker analysis).
* • ISUP Grade 1(Gleason 3+3) and Grade 2 (Gleason 3+4) and Grade 1 (Gleason 3+3, with PSA≥10, or stage ≥ T2b)
* Estimated life expectancy is ≥ 10 years
* Candidate for primary curative therapy (Radical prostatectomy or radiation) if cancer progresses.
* Tolerated previous transrectal ultrasound guided biopsy procedure under local anesthetic

  * Uncomplicated previous TRUS biopsy procedure (i.e., no prior hospitalization due to sepsis, prostatic abscess or severe hemorrhage following TRUS prostate biopsy)
* Willing to undergo the intratumoral (IT) injection of the Poly-ICLC into the prostatic tumor as per the protocol
* No prior hormonal therapy with exception of with the exception of oral 5-alpha-reductase inhibitors (finasteride, dutasteride, etc.). Subjects should be off the medication ≥ 6 months from screening
* No prior radiation therapy (external beam or brachytherapy) to the pelvis or prostate.
* No clinically significant infections as judged by the treating investigator.
* No characteristics suggesting a potential higher risk of infection with intraprostatic injections:

  * Recurrent urinary tract infections or history of prostatitis within 3 months prior to enrollment into the study.
  * Urine analysis positive for nitrites and leucocyte esterase. Such subjects could be considered for the study after treatment and resolution of the infection.
  * Active proctitis
  * History of prostatic abscess
  * Taking immunosuppressive medication including systemic corticosteroids
  * Active hematologic malignancy
* No uncontrolled angina, congestive heart failure or MI within 6 months.
* Subjects with history of HIV (if CD4+ T cell counts are ≥350 cells/μL on established ART therapy), Hepatitis B (with viral load below limits of quantification) or Hepatitis C (who have completed a curative therapy and have a viral load below the limit of quantification) are eligible for this study.
* No treatment with any investigational agent for any medical condition within 28 days prior to being registered for protocol therapy.
* Patients with the potential for impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Contraception must be continued for at least 2 months following the last dose of poly-ICLC. While animal reproductive studies have been negative, the simulated viral infection and anti-proliferative activity of this experimental drug may theoretically affect the developing fetus or nursing infant.
* Adequate end organ function as determined by the following laboratory values:

  * White blood cell count (WBC) ≥ 2.5 k/mm^3
  * Absolute neutrophil count (ANC) ≥ 1.5 k/mm^3
  * Hemoglobin (Hgb) ≥ 8.0 g/dL
  * Platelets ≥ 100 k/mm^3
  * Calculated creatinine clearance of > 60 cc/min using the Cockcroft-Gault formula:
  * Males: [(140 - Age in years) × Actual Body Weight in kg]/[72 × Serum Creatinine (mg/dL)]
  * Bilirubin ≤ 2.0 x ULN
  * Aspartate aminotransferase (AST) ≤ 2.5 x ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN

Exclusion Criteria:

* Received local or systemic curative therapy for prostate cancer
* Subjects with neuroendocrine tumors
* ISUP Gleason Grade Group (>3), or Gleason 3+3 plus PSA ≤ 10 or Stage ≤T2a
* Evidence of locally advanced disease
* Subject has evidence of any other malignancy
* Allergy to any antibiotics, as IT administration requires prophylactic antibiotics.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 114 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects without Gleason group upgrade after treatment | at 12 months
  Proportion of subjects without Gleason group upgrade after treatment with Poly-ICLC or control, as determined by histological examination of prostate biopsy at the one year time point.
Proportion of subjects without Gleason group upgrade after treatment | at 36 months
  Proportion of subjects without Gleason group upgrade after treatment with Poly-ICLC or control, as determined by histological examination of prostate biopsy at the three years time point.
Proportion of subjects without Gleason group downgrade after treatment | at 12 months
  Proportion of subjects with Gleason group downgrade after treatment with Poly-ICLC or control, as determined by histological examination of prostate biopsy at the one year time point.
Proportion of subjects without Gleason group downgrade after treatment | at 36 months
  Proportion of subjects with Gleason group downgrade after treatment with Poly-ICLC or control, as determined by histological examination of prostate biopsy at the 3 years time point.

SECONDARY OUTCOMES:
Number of subjects who experience adverse events per NCI-CTCAE 5.0 | At 12 months
  The number of subjects who experience adverse events, and/or dose-limiting toxicities (DLT) as defined by common criteria developed by the United States National Institutes of Health (NIH), National Cancer Institute and put forward as the Common Terminology Criteria for Adverse Events (NCI-CTCAE 5.0).
Number of subjects who experience adverse events per NCI-CTCAE 5.0 | At 36 months
  The number of subjects who experience adverse events, and/or dose-limiting toxicities (DLT) as defined by common criteria developed by the United States National Institutes of Health (NIH), National Cancer Institute and put forward as the Common Terminology Criteria for Adverse Events (NCI-CTCAE 5.0).
Number of subjects who receive prostate cancer treatment | At 12 months
  Number of subjects who receive prostate cancer treatment (e.g. surgery, radiation, hormone therapy)
Number of subjects who receive prostate cancer treatment | At 36 months
  Number of subjects who receive prostate cancer treatment (e.g. surgery, radiation, hormone therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Sujit S Nair, PhD, Study Director — Assistant Professor and Director of GU Immunotherapy Research; Dimple Chakravarty, PhD, Study Director — Assistant Professor
Locations (1):
- Icahn School of Medicine at Mount Sinai (ISMMS), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Proposals should be directed to monali.fatterpekar@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link tbd).